CLINICAL TRIAL: NCT03852511
Title: A Multicentre, Open Label, Non-randomised First in Human Study of NG-350A (Monotherapy), and NG-350A With a Check Point Inhibitor in Patients With Metastatic or Advanced Epithelial Tumours
Brief Title: First in Human Study of NG-350A (an Oncolytic Adenoviral Vector Which Expresses an Anti-CD40 Antibody)
Acronym: FORTITUDE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Akamis Bio (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NG-350A-01
Record Dates: First submitted 2019-02-11; First posted 2019-02-25 (Actual); Last update posted 2022-06-24 (Actual); Status verified 2022-06

CONDITIONS: Metastatic Cancer; Epithelial Tumor
Keywords: metastatic; epithelial; virus; advanced
MeSH Terms: conditions — Neoplasm Metastasis; Carcinoma; Virus Diseases

STUDY DESIGN:
Intervention Model Description: Patients in Part A will receive a single cycle of NG-350A study treatment, with three single doses on Days 1, 3 and 5 by IV infusion.
  Patients in Part B will receive a single cycle of NG-350A study treatment, with three single doses on Days 1, 3 and 5 by IV infusion, followed by up to 8 cycles of a check point inhibitor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intravenous (Experimental): Patients will receive three single doses of NG-350A by IV infusion, followed by multiple cycles of check point inhibitor treatment.
  Interventions: Biological: NG-350A

INTERVENTIONS:
Biological: NG-350A — NG-350A is oncolytic adenoviral vector which expresses a full length agonist anti-CD40 antibody at the site of virus replication.

SUMMARY:
This study will evaluate the safety, tolerability and preliminary efficacy and also pharmacokinetics, immunogenicity and other pharmacodynamic effects to elucidate the mechanism of action of NG-350A, either alone or in combination with a check point inhibitor, in patients with advanced or metastatic epithelial tumours.

DETAILED DESCRIPTION:
Phase Ia of this study is a dose escalation phase, investigating NG-350A administration by intravenous (IV) infusion, either alone or in combination with a check point inhibitor. Phase Ib of this study comprises of a Combination Dose Efficacy Expansion with NG-350A in combination with a check point inhibitor.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent to participate
2. Aged 18 years or over
3. Have one of eleven histologically or cytologically confirmed metastatic or advanced carcinomas or adenocarcinomas that have progressed after at least one line of systemic therapy and are incurable by local therapy

   a. Tumour types eligible are: UC, SCCHN, MSI high/dMMR cancer, NSCLC, uterine/endometrial cancer, cervical cancer, oesophageal cancer, gastric cancer, cutaneous squamous cell carcinoma, HCC and TNBC
4. Additional tumour type specific criteria:

   1. UC: carcinoma of the renal pelvis, ureter, bladder, or urethra that showed predominantly transitional-cell features on histologic testing
   2. SCCHN with oropharyngeal cancer: known HPV p16 status
   3. MSI-high/dMMR cancer: MSI-high/dMMR status must be confirmed by an approved test
   4. NSCLC: either squamous or non-squamous histology
   5. Gastric cancer: gastric or gastroesophageal junction adenocarcinoma
5. All patients enrolled in combination therapy cohorts with check point inhibitor (dose escalation and efficacy expansion phases) must have received prior treatment with a PD 1/PD-L1 inhibitor therapy (prior PD-1/PD-L1 may have been given as monotherapy or combination therapy)

   1. In combination dose-escalation, patients may have received a PD 1/PD L1 inhibitor as part of any prior line of therapy (additional criteria apply when this is the most recent line of therapy - see below)
   2. In dose expansion cohorts, patients must have been treated with a PD 1/PD-L1 inhibitor as part of their most recent treatment
   3. For all patients who received PD-1/PD-L1 inhibitor therapy as part of their most recent line of treatment (includes dose-escalation and all patients in dose-expansion), this must have been for a minimum of 6 weeks and maximum of 6 months, with best response of SD or PD - Patients with PD following treatment with a PD-1/PD-L1 inhibitor as their most recent therapy must have a <50% increase in disease burden
6. At least one measurable site of disease according to RECIST Version 1.1 criteria; this lesion must be either (i) outside a previously irradiated area or (ii) progressive if it is in a previously irradiated area
7. Tumour accessible for biopsy, biopsy deemed safe for biopsy by the Investigator, and patient willing to consent to tumour biopsies
8. Ability to comply with study procedures in the Investigator's opinion
9. Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
10. Predicted life expectancy of 6 months or more
11. Adequate lung reserve
12. Adequate renal function
13. Adequate hepatic function
14. Adequate bone marrow function
15. Coagulation profile within the normal range (international normalized ratio ≤1.5)
16. Meeting reproductive status requirements

Exclusion Criteria:

1. Prior or planned allogeneic or autologous bone marrow or organ transplantation
2. Splenectomy
3. Active infections requiring antibiotics, physician monitoring or systemic therapy within 1 week of the anticipated first dose of study drug, or recurrent fevers (>38.0˚C) associated with a clinical diagnosis of active infection
4. Active viral disease or positive test for hepatitis B virus using hepatitis B surface antigen test or positive test for hepatitis C virus (HCV) using HCV ribonucleic acid (RNA) or HCV antibody test indicating acute or chronic infection. Positive test for HIV or AIDS
5. Patients who have active autoimmune disease that has required systemic therapy in the past 2 years, are immunocompromised in the opinion of the Investigator, or are receiving systemic immunosuppressive treatment

   a. Patients with vitiligo, type I diabetes mellitus, asthma/atopy, residual hypothyroidism due to autoimmune disease (which only requires hormone replacement therapy), or conditions not expected to recur in the absence of an external trigger are permitted to enrol providing they comply with the other eligibility criteria relating to renal function. Use of inhaled corticosteroids, local steroid injection, or steroid eye drops is allowed
6. Treatment with any live, live attenuated or COVID-19 vaccine in the 28 days before the first dose of NG 350A

   a. COVID-19 vaccines known not to be based on an adenoviral vector (e.g. mRNA vaccines) are not subject to the 28-day exclusion (see exclusion criterion 7)
7. Treatment with any other vaccine (including known non-adenoviral COVID-19 vaccines) in the 7 days before first dose of NG-350A
8. History of prior Grade 3-4 acute kidney injury or other clinically significant renal impairment
9. History of clinically significant interstitial lung disease or non-infectious pneumonitis
10. Lymphangitic carcinomatosis (clinically suspected or radiographic evidence)
11. Infectious or inflammatory bowel disease in the 3 months before the first dose of study treatment
12. Myocardial infarction, stroke or other significant cardiovascular or cerebrovascular event in the 12 months before the first dose of study treatment
13. Pulmonary embolism, deep vein thrombosis, or other uncontrolled thromboembolic event in the 12 months before the first dose of study treatment, or current treatment with therapeutic or prophylactic anticoagulation therapy
14. Grade 3 or 4 gastrointestinal bleeding (or risk factors for gastrointestinal bleeding) or haemoptysis in the 3 months before first dose of study treatment, or any history of bleeding requiring an investigative procedure (e.g. endoscopy), transfusion or hospitalisation in the 12 months before the first dose of study treatment
15. Tumour location/extent considered by the Investigator to present a significant risk if tumour flare or necrosis were to occur (e.g. an initial increase in tumour size that may lead to intestinal, airway or ureter obstruction, or penetrating tumour infiltration of major blood vessels, or other hollow organs potentially at risk of perforation)
16. Use of the following prior therapies/treatments:

    1. Treatment with any other anti CD40 antibody at any time
    2. Treatment with an investigational or licensed anti-cancer monoclonal antibody (mAb), immune checkpoint inhibitor, immune stimulatory treatment or other biological therapy in the 28 days prior to the first dose of study treatment. Prior anti PD-1 / PD-L1 therapy is permitted without a 'washout' phase
    3. Treatment with an investigational or licensed chemotherapy, targeted small molecule or other investigational drug in the 14 days or five half-lives (whichever is shorter) before the first dose of study treatment
    4. Major surgery in the 28 days before the first dose of study treatment or radiation therapy in the 14 days before the first dose of study treatment

    i. Bisphosphonate therapy or treatment with Receptor Activator of Nuclear factor Kappa-B (RANK)-ligand inhibitors for metastatic bone disease is permitted
17. All toxicities attributed to prior anti-cancer therapy (including radiation therapy) other than alopecia must have resolved to Grade 1 or baseline before the first dose of study treatment. Patients with toxicities (other than renal toxicities) attributed to prior anti-cancer therapy that are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum-based therapy, are permitted to enrol
18. Treatment with the antiviral agents ribavirin, adefovir, lamivudine or cidofovir within 7 days prior to the first dose of study treatment; or pegylated interferon (PEG-IFN) in the 14 days before the first dose of study treatment
19. Known allergy/immune-related adverse reactions to NG-350A transgene or immune checkpoint inhibitor products or formulation; severe hypersensitivity to another monoclonal antibody
20. Other prior malignancy active within the previous 3 years, except for local or organ confined early-stage cancer that has been definitively treated with curative intent, does not require ongoing treatment, has no evidence of residual disease and has a negligible risk of recurrence and is therefore unlikely to interfere with the primary and secondary endpoints of the study, including response rate and safety
21. Symptomatic brain metastases or any leptomeningeal metastases that are symptomatic and/or require treatment. Patients with brain metastases are eligible if these have been treated (surgery, radiotherapy). Both surgery and or radiotherapy must have been completed at least 2 weeks before first dose of study treatment. There must also be no requirement for immunosuppressive doses of systemic corticosteroids (>10 mg/day prednisone equivalent) for at least 2 weeks before the first dose of study treatment
22. Any serious or uncontrolled medical disorder that, in the opinion of the Investigator or the Medical Monitor, may increase the risk associated with study participation or study treatment administration, impair the ability of the patient to receive protocol therapy or interfere with the interpretation of study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events, serious adverse events, adverse events meeting protocol-defined DLT criteria, severe adverse events, adverse events leading to study treatment or study discontinuation, and adverse events resulting in death. | Throughout study to end of study treatment visit (Week 24 or +30 days after last study drug dose)
  Characterise the safety and tolerability of NG-350A, in combination with a check point inhibitor, by reviewing reported Adverse Events (AEs) and Serious Adverse Events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Aung Naing, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (5):
- United States (5):
  - University of California, Los Angeles (UCLA), Santa Monica, California
  - University of Colorado, Aurora, Colorado
  - Memorial Sloan Kettering Cancer Center (MSKCC), New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Khalil DN, Prieto Gonzalez-Albo I, Rosen L, Lillie T, Stacey A, Parfitt L, Soff GA. A tumor-selective adenoviral vector platform induces transient antiphospholipid antibodies, without increased risk of thrombosis, in phase 1 clinical studies. Invest New Drugs. 2023 Apr;41(2):317-323. doi: 10.1007/s10637-023-01345-8. Epub 2023 Mar 10. PMID 36897458